CLINICAL TRIAL: NCT03225703
Title: The Effect of High Impact Exercise on Bone and Articular Cartilage in Post-menopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Katherine Brooke-Wavell, Senior Lecturer in Human Biology, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R16-P149
Record Dates: First submitted 2017-04-05; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Osteoporosis, Postmenopausal; Osteoarthritis, Knee; BMD
Keywords: Exercise; Osteoporosis; Osteoarthritis; MRI; DXA; High Impact; Cartilage; Bone
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoarthritis, Knee; Motor Activity; Osteoporosis; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Participants will complete a unilateral exercise intervention and be randomly assigned an exercise leg. This allows for internal control, non exercise leg. The exercise and control leg will be analysed for significant differences following completion of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Leg (Active Comparator): Left or right leg randomly assigned as exercise leg in a unilateral, exercise intervention. This will be a progressive exercise programme with the aim being to complete 50 multidirectional hops completed daily. (Hopping)
  Interventions: Behavioral: Hopping
- Non exercise Leg (No Intervention): Randomly assigned non-exercise, control leg.

INTERVENTIONS:
Behavioral: Hopping — A unilateral, hopping based exercise programme lasting six months.
  Arms: Exercise Leg

SUMMARY:
Osteoarthritis (OA) and osteoporosis (OP) affect large numbers of the population. Around 8 million people in the UK are affected by OA and over 300,000 people present with fragility fractures in the UK each year. High impact exercise has been shown to improve markers of bone health but the effect of this exercise on the cartilage is less well understood. A six month, one leg, exercise program based on hopping will be carried out by a group of post-menopausal women. Post-menopausal women are particularly at risk from OP and the research should give information on the feasibility of this type of exercise program in this age group and the effect on cartilage. Participants will be aged between 55 and 70 (at least five years post menopause) with no conditions that would limit their ability to complete the exercise program.

To assess changes in participants' cartilage and bone properties they will be asked to attend several meetings at Loughborough University. Before and after the exercise program participants will have bone density scans and MRI scans of the knee joint. A subset (n=4) will undergo high resolution bone scans that can demonstrate changes in bone structure. The intervention is a home based exercise programme lasting approximately 10 minutes per day. Initially this will be individualised to each participant with the end goal being daily exercise sessions. The programme will last for six months with supervised sessions offered throughout the trial. Using an intervention affecting just one leg will allow the research team to use the other leg as a control.

The research team hypothesise that in a population of post-menopausal women, a six month, unilateral exercise intervention will improve bone mineral density at the proximal femur with no negative effects on articular cartilage.

DETAILED DESCRIPTION:
The research is a 6 month, intervention study of unilateral (single limb) exercise with the changes in a randomly chosen exercise leg being compared to those in the other (control) leg.

Potential participants (women aged 55-70) will be approached via existing links in the community, at local community centres, through local media, posters and flyers. After initial contact to determine whether they meet the inclusion/exclusion criteria they will be invited to join the study and sent the participant information sheet (PIS). If they then wish to aid in the research they will be invited to a first meeting at Loughborough University.

At the initial meeting the participant can further discuss the project and PIS with the research team. If they fully understand the project and are happy to take part they will be invited to sign the informed consent form. At this stage each participant will be anonymised using a project code. Screening and baseline measurements will then be taken.

Screening questionnaires will be taken following consent to the study. These include a demographic questionnaire, health screen questionnaire, calcium intake questionnaire, physical activity readiness questionnaire (PAR-Q) and bone physical activity questionnaire (BPAQ).

Dual X-ray Absorptiometry (DXA) scans of the whole body, anterior-posterior (AP) spine and dual femur will be taken for each participant to give baseline measurements of bone mineral density.Standard positioning procedures for the measurement being taken will be utilised to allow the calculation of the T-score.

Functional tests will be performed to investigate hopping and balance ability. Unilateral balance will be analysed by measuring postural sway using a force platform. Participants will be asked to balance on one leg for up to 30 seconds. Amplitude of displacement will be calculated, this is the distance between the maximum and minimum centre of pressure (COP) in both directions. COP path length is the total distance travelled and will be calculated and divided by the trial time to give the COP velocity.

Maximal hop height will be measured by recording the vertical displacement of a marker placed on the lumbar spine of each participant whilst conducting a maximal hop. This will be repeated for each leg. The ground reaction force (GRF) of the maximal hop will be recorded using a force platform. Participants will be asked to remain still on the platform for 5 seconds to determine body weight. From this position participants will be asked to lift one leg from the platform and perform a counter movement, maximal hop using their arms to help with propulsion and ensure maximal hop height. After one or two familiarisation attempts the participant will be asked to complete three maximal hops. Allowing for repeats if they do not land fully on the force platform. The peak GRF recorded from these three attempts will be used in the final analysis.

Ground reaction forces during a set of ten hops, which is the end goal of the exercise programme, will be recorded on a force platform. Participants will be asked to remain still on the platform for 5 seconds to determine body weight. From this position participants will be asked to lift one leg from the platform and perform ten counter movement hops using their arms to help with propulsion if able. At the baseline measurements participants will be asked to perform ten hops to the best of their ability, with a rigid support available for them to lean on

A second appointment will be arranged to acquire baseline MRI scans of each knee joint. This will involve the safety checks, conversation with the radiographers and scan times of up to one hour.

Following the MRI scans the exercise leg will be randomly assigned using opaque envelopes. Each envelope will contain a note saying either 'left leg' or 'right leg'. The envelopes will be split into smaller subgroups of eight for minimisation. This will remove the possibility of the first half of volunteers choosing the same leg and removing the randomisation effect on the second half. Participants will be presented with a training diary and instructions on how to complete the exercise programme over six months. The first day of exercise will be completed with the research team at this appointment and the intervention considered started. This second meeting should last for approximately 90 minutes.

The required exercise lasts for no longer than 10 minutes each session and can be performed at home. The intervention will be personalised to the individual's ability and the frequency of the exercise will steadily increase as the participant improves, until the exercise is completed daily. Regular group sessions at Loughborough University will be offered to all participants. The exercise time will remain at ten minutes but the session will be longer, allowing for discussion and check-ups with participants. These will be weekly sessions for the first two months and then once a month for the remaining time.

Follow up measurements will take place six months after the commencement of the exercise programme. Repeat DXA, MRI and functional outcome tests will be carried out on all participants, following the same protocol as at baseline. Again this will occur over two meetings at Loughborough University.

A subset (n=4) will undergo high resolution bone scans (HR-pQCT) that can demonstrate changes in bone structure. This measurement will be taken at the distal tibia and lasts around three minutes per leg. Measurements will be taken pre and post the six month exercise intervention.

Descriptive statistics will be calculated to give information on mean values and variation (standard deviation) of the cohort. This will include age, height, body mass, BMI and time since last menstruation.

Using Levene's test when comparing the exercise to control leg and Mauchly's test of sphericity to compare from baseline to end of study, the variance of the data will be analysed. Normal distribution will be analysed using Shapiro-Wilks test and visual examination of Q-Q plot. If variance is shown to be homogenous and distribution normal within the population then a repeated measures analysis of variance (RM-ANOVA)will be used to detect any significant differences between leg (exercise versus control, time (baseline versus post-intervention) or leg x time interaction in the outcome variable described previously. If any of the outcome measures do not meet the assumptions to conduct parametric tests i.e. ANOVA then Kruskal-Wallis H test will be used to detect any significant change in differences.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal - at least 12 months since last menstruation and/or hysterectomy, oophorectomy or hormonal contraceptive use

Exclusion Criteria:

* Existing knee, hip or back injury.
* Any medical conditions or injuries which exclude participation in an exercise intervention e.g. heart conditions, hypertension
* BMI > 30 kg/m2
* Participation in a study involving ionising radiation in the previous 12 months.
* Exercise involving ground reaction forces greater than that of jogging more than once a week.
* Contraindications to MRI or DXA
* Osteoporotic (FRAX score requiring the participant is advised to seek treatment)
* Medication affecting bone metabolism or density

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Change in T2 Relaxation Time (ms) | 6 months (pre and post intervention)
  T2 mapping is an indicator of the water content in cartilage, with longer relaxation times a marker of cartilage degeneration

SECONDARY OUTCOMES:
Change in Femoral neck bone mineral density (g/cm2) | 6 months (pre and post intervention)
Change in Femoral neck bone mineral content (g) | 6 months (pre and post intervention)
Change in Spine bone mineral density (g/cm2) | 6 months (pre and post intervention)
Change in Spine bone mineral content (g) | 6 months (pre and post intervention)
Change in Postural sway (mm) | 6 months (pre and post intervention)
Change in Maximal hop height (mm) | 6 months (pre and post intervention)
Change in Ground Reaction force Maximal Hop (N) | 6 months (pre and post intervention)
Change in Ground Reaction force for a set of ten hops (N) | 6 months (pre and post intervention)
Change in BMD(D100) (mg HA/cm3) | 6 months (pre and post intervention)
  Volumetric Bone mineral density
Change in Total bone mass (mg) | 6 months (pre and post intervention)
Change in BV/TV (%) | 6 months (pre and post intervention)
  Percent bone volume
Change in pBV/TV (%) | 6 months (pre and post intervention)
  Plate bone volume fraction
Change in rBV/TV (%) | 6 months (pre and post intervention)
  Rod bone volume fraction
Change in pBV/rBV (%) | 6 months (pre and post intervention)
  Plate to - rod ratio
Change in pBV/BV (%) | 6 months (pre and post intervention)
  Plate tissue fraction
Change in rBV/BV (%) | 6 months (pre and post intervention)
  Rod tissue fraction
Change in Bone surface(BS) (mm2) | 6 months (pre and post intervention)
Change in BS/TV (mm-1) | 6 months (pre and post intervention)
  Bone surface density
Change in Tb.Th (mm) | 6 months (pre and post intervention)
  Trabecular thickness
Change in Tb.Sp (mm) | 6 months (pre and post intervention)
  Trabecular Separation
Change in Tb.N (mm-1) | 6 months (pre and post intervention)
  Trabecular number
Change in Tb.Pf | 6 months (pre and post intervention)
  Trabecular bone pattern (Tb.PF) follows the course of stress lines in the bone. This measurement indicates where the bone is under increased stress.
Change in Conn.D (mm-3) | 6 months (pre and post intervention)
  Connectivity density
Change in DA | 6 months (pre and post intervention)
  Degree of anisotropy
Change in τ | 6 months (pre and post intervention)
  Tortuosity (τ) is a measure of how well a structure can curve and bend easily. This is an indicator of where the most stress is on the bone structure.
Change in SMI | 6 months (pre and post intervention)
  Structural model index
Change in BRV (mm3) | 6 months (pre and post intervention)
  Bone resorption volume
Change in BFV (mm3) | 6 months (pre and post intervention)
  Bone formation volume
Change in BRM (mg) | 6 months (pre and post intervention)
  Bone resorption mass
Change in BFM (mg) | 6 months (pre and post intervention)
  Bone formation mass
Change in BRF (%) | 6 months (pre and post intervention)
  Bone resorption fraction
Change in BFF(%) | 6 months (pre and post intervention)
  Bone formation fraction
Change in BRR(mm3/week) | 6 months (pre and post intervention)
  Bone resorption rate
Change in BFR(mm3/week) | 6 months (pre and post intervention)
  Bone formation rate
Change in Trabecular orientation distribution (Tb.O.D) (angle in degrees) | 6 months (pre and post intervention)
  This is a measurement of the orientation of the trabeculae in the distal tibia relative to the central axis tibial shaft. The orientation can be categorised into transvers direction and longitudinal direction along the tibial shaft
Change in Ct.Th(mm) | 6 months (pre and post intervention)
  Cortical thickness
Change in B.Po(%) | 6 months (pre and post intervention)
  Bone porosity
Change in Po.Dm(mm) | 6 months (pre and post intervention)
  Pore diameter
Change in Pore volume distribution | 6 months (pre and post intervention)
Change in Failure load (N) | 6 months (pre and post intervention)
Change in Strain | 6 months (pre and post intervention)
  This analyses the change in length of the bone over the time period, expressed as % change.
Change in Stiffness (N/mm) | 6 months (pre and post intervention)
Change in Young's Modulus (GPa) | 6 months (pre and post intervention)
Change in Mechanical anisotropic ratio | 6 months (pre and post intervention)
Change in Strain energy density (J/m3) | 6 months (pre and post intervention)
Change in Strain gradient (με/mm) | 6 months (pre and post intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Brooke-Wavel, PhD, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to have scans available on a public database.

REFERENCES:
- [Derived] Du J, Hartley C, Brooke-Wavell K, Paggiosi MA, Walsh JS, Li S, Silberschmidt VV. High-impact exercise stimulated localised adaptation of microarchitecture across distal tibia in postmenopausal women. Osteoporos Int. 2021 May;32(5):907-919. doi: 10.1007/s00198-020-05714-4. Epub 2020 Nov 16. PMID 33196852